CLINICAL TRIAL: NCT03556423
Title: Pain in Individuals With Knee Osteoarthritis : Beyond the Joint and the Musculoskeletal System
Brief Title: Neurophysiological Mechanisms Involved in Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Guillaume Léonard, Professor, Université de Sherbrooke
Other Study IDs: 2015-454-IUGS
Record Dates: First submitted 2018-05-16; First posted 2018-06-14 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Knee Osteoarthritis; Chronic Pain
Keywords: Arthritis; Chronic pain; Transcranial magnetic stimulation (TMS); Magnetic resonance imaging (MRI); Conditioned pain modulation (CPM); Clinical measures; Knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Chronic Pain; Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Introduction: Total knee arthroplasty (TKA) is an effective intervention to relieve people with osteoarthritis (OA). Nevertheless, 15 to 30% of patients continue to experience severe pain following surgery. Recent data suggest that central nervous system (CNS) changes may play a role in OA pain and possibly explain why some patients have poorer clinical outcomes following TKA. Objectives: Our main objectives are to explore the relationship between OA pain and (1) the integrity of corticospinal system, (2) the efficacy of descending pain inhibition circuits. Methods: Fifty-two patients waiting for TKA will be recruited. The integrity of the corticospinal projections will be measured using transcranial magnetic stimulation (recruitment curve of the affected quadriceps femoris muscle) and the descending pain inhibition circuits (bulbospinal projections) will be assessed by a counter-irritation paradigm (i.e., conditioned pain modulation with immersion of the arm in painfully cold water). Diffuse tension imaging (DTI) will also be used to quantify the strength of these corticospinal and bulbospinal projections. Clinical outcomes will be evaluated before and after arthroplasty with a series of validated questionnaires such as the WOMAC Scale, the McGill Pain Questionnaire and the Brief Pain Inventory. These different neurophysiological and clinical measures will be taken before surgery, 6 months after surgery and 1 year post-surgery. Anticipated results: The investigators expect a moderate association between pain and the strength of the corticospinal and bulbospinal projections. Moreover, it is expected that there will be a moderate association between the strength of the corticospinal/bulbospinal projections and the clinical evolution of patients.

DETAILED DESCRIPTION:
See outcome measures

ELIGIBILITY:
Inclusion Criteria:

* Being an adults aged 50-79 years old with a diagnosis of knee OA and waiting for a primary arthroplasty
* Refrain from consuming cigarettes and caffeine 2 hours and 6 hours before testing, respectively
* Refrain from taking short-acting analgesics (e.g., acetaminophen) 6 hours before testing

Exclusion Criteria:

* Having difficulty understanding french language
* Having a diagnosis of neurological disorder or diagnosis of chronic pain (other knee OA)
* Having metal implants in the skull
* Having pacemaker or neurostimulator
* Being pregnant
* Being epileptic

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 50-79 years old with a diagnosis of knee OA and waiting for a primary arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline - Integrity of the corticospinal system | Before surgery, 6 months and 1 year post-surgery
  This outcome will be measured by transcranial magnetic stimulation (TMS)
Change from baseline - Descending pain inhibition circuits | Before surgery, 6 months and 1 year post-surgery
  This outcome will be measured by a counter-irritation paradigm (conditioned pain modulation using a thermode and a bath of circulating cold water)
Change from baseline - Pain intensity | Before surgery, 6 months and 1 year post-surgery
  This outcome will be measured by a visual analogue scale (VAS). The VAS is a straight horizontal line of fixed length, usually 10 cm. The ends are defined as the extreme limits of the parameter to be measured; 0 = "no pain", 10 = "the worst imaginable pain". Using a ruler, the score is determined by measuring the distance (cm) on the 10 cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-10. A higher score indicates greater pain intensity.
Change from baseline - Pain, stiffness and physical function | Before surgery, 6 months and 1 year post-surgery
  This outcome will be measured by Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)

SECONDARY OUTCOMES:
Pain catastrophizing | Before surgery, 6 months and 1 year post-surgery
  This outcome will be measured with the Pain Catastrophizing Scale (PCS) . The PCS inquire participants to reflect on past painful experiences, and to indicate the degree to which they experienced each of 13 thoughts or feelings when experiencing pain. Each item of the PCS is scored on a 5-point scale where 0 = not at all and 4 = all the time. PCS yields three subscale scores assessing rumination, magnification and helplessness. The PCS total score is computed by summing responses to all 13 items. The PCS yields a total score ranging from 0 to 52. Higher values on this scale represent a greater tendency of the subject to perceive pain negatively and to foresee the consequences of pain in a more catastrophic way.
Kinesiophobia | Before surgery, 6 months and 1 year post-surgery
  This outcome will be measured with the Tampa Scale of Kinesiophobia (TSK) . The TSK is a 17-item self-report checklist using a 4-point Likert scale that was developed as a measure of fear of movement or (re)injury. The total score ranges between 17 and 68. A high value on the TSK indicates a high degree of kinesiophobia, and a cutoff score was developed by Vlaeyen (1995), where a score of 37 or over is considered as a high score, while scores below that are considered as low scores.
Anxiety | Before surgery, 6 months and 1 year post-surgery
  This outcome will be measured with the Spielberger's State-Trait Anxiety Inventory
Qualitative aspect of pain | Before surgery, 6 months and 1 year post-surgery
  This outcome will be measured by the McGill Pain Questionnaire
Impact of pain on physical function and quality of life | Before surgery, 6 months and 1 year post-surgery
  This outcome will be measured by the Brief Pain Inventory (BPI)
Functional autonomy, social autonomy | Before surgery, 6 months and 1 year post-surgery
  This outcome will be measured by the SMAF questionnaire

OTHER OUTCOMES:
Level of physical activity | Before surgery, 6 months and 1 year post-surgery
  Physical Activity Scale for the Elderly (PASE)
Hypersensitivity of central nervous system | Before surgery, 6 months and 1 year post-surgery
  This outcome will be measured by the Central Sensitization Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Leonard, Ph.D., pht., Principal Investigator — Centre de Recherche sur le Vieillissement (CdRV)
Locations (2):
- Canada (2):
  - Centre de recherche sur le vieillissement (CdRV), Sherbrooke, Quebec
  - CRCHUS: Centre de recherche du centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Undecided